CLINICAL TRIAL: NCT07364617
Title: Fecal Microbiota Transplantation for the Treatment of Steroid Refractory Acute Gastrointestinal Graft-Versus-Host Disease in Patients After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Fecal Microbiota Transplantation for Steroid-Refractory Acute GI GVHD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Hsiaowen Kao, M.D., Division of Hematology-Oncology, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202401777A0; LK20250520001 (Other Grant/Funding Number: Chang Gung Medical Foundation)
Record Dates: First submitted 2025-12-02; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Graft vs Host Disease
Keywords: Acute Gastrointestinal Graft-versus-Host Disease; fecal microbiota transplantation; steroid-refractory
MeSH Terms: conditions — Graft vs Host Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This prospective, single-arm, open-label phase II study evaluates fecal microbiota transplantation (FMT) as treatment for adults with steroid-refractory stage II-IV acute gastrointestinal graft-versus-host disease (GI-GvHD) after allogeneic hematopoietic stem cell transplantation. Participants receive 250 mL microbiota fluid delivered to the terminal ileum/cecum via ileocolonoscopy or to the duodenum via panendoscopy, with a second FMT given 7-21 days later and an optional third dose based on response. The study assesses event-free survival, overall and complete response rates at Days 28 and 56, steroid reduction, relapse, survival, and safety including infections and procedure-related complications. Serial clinical, microbiologic, and immunologic evaluations are performed to characterize treatment effects and adverse events. Total planned enrollment is 35 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Participants receive 250 mL microbiota fluid delivered to the terminal ileum/cecum via ileocolonoscopy or to the duodenum via panendoscopy, with a second FMT given 7-21 days later and an optional third dose based on response.
  Interventions: Biological: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Biological: Fecal microbiota transplantation (FMT) — About 250 mL microbiota fluid, containing approximately 60 cm³ of stool materials; 6x10¹³ bacteria, will be delivered to the terminal ileum/cecum via ileocolonoscopy or to the duodenum via panendoscopy, with a second FMT given 7-21 days later and an optional third dose based on response.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective treatment for various hematologic diseases. However, one of the major challenges of allo-HSCT is the occurrence of graft-versus-host disease (GvHD), particularly acute gastrointestinal GvHD (GI-GvHD). GvHD occurs when donor T cells recognize the recipient's tissue as foreign and mount an immune attack against it. Acute GI-GvHD is a common complication following allo-HSCT and a significant cause of mortality. If the initial steroid treatment for acute GvHD fails, mortality rates can reach as high as 81%.

Recent studies have shown a strong association between reduced gut microbiota diversity and high mortality in patients with acute GI-GvHD, highlighting the critical role of the gut microbiome in regulating immune responses and maintaining intestinal homeostasis. Consequently, fecal microbiota transplantation (FMT) has emerged as a potential therapeutic strategy aimed at restoring a healthy gut microbiome and improving clinical outcomes in patients with acute GI-GvHD.

This study aims to evaluate the efficacy and safety of FMT in patients with steroid-refractory or steroid-resistant acute GI-GvHD. The findings of this research will contribute to establishing FMT as a potential and effective treatment option for managing severe acute GI-GvHD, thereby improving patient outcomes and reducing transplant-related mortality.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, phase II clinical trial evaluating the safety and efficacy of fecal microbiota transplantation (FMT) in adult patients with steroid-refractory acute gastrointestinal graft-versus-host disease (acute GI-GvHD) following allogeneic hematopoietic stem cell transplantation (allo-HSCT). Eligible patients will receive 250 cc microbiota fluid prepared from healthy screened donors, delivered into the terminal ileum or cecum via ileocolonoscopy, or into the terminal duodenum via panendoscopy. The study aims to assess event-free survival, overall and complete response rates, survival outcomes, changes in steroid exposure, adverse events, and microbiological/immunological biomarkers. A total of 35 participants will be enrolled over a planned 2-year study period.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II to IV steroid refractory acute GI-GvHD in allo-HSCT recipients

   1. Stage II to IV acute GI-GVHD subjects, having >1000 mL stool per day, diarrhea > 5 times/day, or abdominal cramping, bleeding or ileus, AND
   2. Resistant to a first-line therapy with corticosteroids (CS)

   <!-- -->

   1. Lack of improvement after 5 days of treatment with CS at 2 mg/kg/d methylprednisolone or other CS with equivalent dose,
   2. Progression after 3 days of treatment with CS at 2 mg/kg/d methylprednisolone or other CS with equivalent dose.
2. Age ≥ 18 years old.
3. Allo-HSCT with any type of donor, stem cell source, GvHD prophylaxis or conditioning regimen.
4. Allow vancomycin-resistant enterococcus (VRE) colonization and asymptomatic cytomegalovirus (CMV) viremia, which is defined as a detectable CMV viral load in plasma but without tissue-invasive disease.
5. Patients able to have a minimum of 12 hours discontinuation of systemic antibiotics in order to perform the allogeneic FMT (antiviral and antifungal agents are allowed)
6. Signature of informed and written consent by the subject or by the subject's legally acceptable representative for patients under guardianship or trusteeship. Subject must understand and voluntarily sign an informed consent form prior to any study-related assessments/procedures being conducted.

Exclusion Criteria:

1. Absolute neutrophil count < 500 cells/uL.
2. Absolute platelet count < 30000 /uL which is not correctable by transfusion
3. Hemodynamically unstable status with the following conditions: systolic blood pressure < 90 mm Hg, pulse oximeter oxygen saturation (SpO2) < 90%, PaO2 < 60 mm Hg, or respiratory rate > 22/minute.
4. Uncontrolled and active infection from bacteria, virus, or fungus as determined by the investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
event-free survival | From first fecal microbiota transplantation to the first event or up to 6 months
overall response rate | on day-28 after first FMT
  at least one stage improvement in acute GI-GvHD
complete response rate | on day-28 after first FMT
  improvement of acute GI-GvHD to stage 0

SECONDARY OUTCOMES:
Overall response rate | on day-56 after first FMT
  at least one stage improvement in acute GI-GvHD
Complete response rate | on day 56 after first FMT
  improvement of acute GI-GvHD to stage 0
Time to response | from the time of first FMT to the time of at least one stage improvement in acute GI-GvHD
Relapse rate | at least two-year follow-up after first FMT
  Relapse defined as at least one stage acute gastrointestinal GvHD progression.
Overall survival | from the time of first FMT to the time of death.
Non-relapse mortality | at least two-year follow-up after first FMT
  death without prior acute gastrointestinal GvHD relapse
Incidence of adverse events | at least two-year follow-up after first FMT
  adverse events include but not limited to infection, cytopenia, viral reactivation, gastrointestinal bleeding, bowel rupture

OTHER OUTCOMES:
Incidence of changes in severity of endoscopic abnormalities and/or histologic evidence of acute GI GVHD relative to baseline assessment. | on second or third FMT
  Gastrointestinal mucosa improvement observed by ileocolonoscopy or panendoscopy findings, or histopathology findings from gastrointestinal tract biopsy
Changes in GvHD related biomarkers | on day-28 after first FMT

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Wen KAO, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The study team plans to share de-identified individual participant data (IPD), including clinical outcomes, laboratory results, and response assessments related to fecal microbiota transplantation for acute GI-GvHD. IPD will be made available after publication of the primary results and following completion of all planned analyses. Data will be shared in a de-identified, password-protected format and will be accessible upon reasonable request to the principal investigator through a formal data-sharing agreement specifying intended use, data protection measures, and prohibition of re-identification. Supporting documents (such as the protocol and statistical analysis plan) may also be available upon request. No public repository upload is currently planned.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting documents (such as the study protocol and statistical analysis plan) will be available starting 12 months after publication of the primary study results. Data will remain available for 5 years after that date. Access will be provided upon reasonable request through a data-sharing agreement with the principal investigator.
Access Criteria: De-identified individual participant data and supporting documents (including the protocol and statistical analysis plan) will be accessible to qualified researchers, academic investigators, research organizations, and regulatory authorities that submit a methodologically sound proposal aligned with the study's scientific objectives. Approved requestors will gain access after signing a data-sharing agreement specifying data-use restrictions, data-security requirements, and a prohibition on re-identification. Data will be shared in a secure, password-protected electronic format provided directly by the study team.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Protocol synopsis 20251219 version 2.1 (2025-12-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT07364617/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Procotoal synopsis english version 2_2 January 14 2026 (2026-01-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT07364617/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol synopsis 20250930 version 2 (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT07364617/Prot_SAP_002.pdf